CLINICAL TRIAL: NCT04957667
Title: Scintigraphic Defecography for Evaluation of Functional Outcome in an Adult Hirschsprung Population
Status: Completed | Type: Observational
Sponsor: University of Southern Denmark (Other)
Responsible Party: Sponsor
Other Study IDs: HD-NQ-2018
Record Dates: First submitted 2021-05-31; First posted 2021-07-12 (Actual); Last update posted 2022-11-09 (Actual); Status verified 2022-11

CONDITIONS: Hirschsprung Disease
Keywords: Hirschsprung disease; Scintigraphic defecography
MeSH Terms: conditions — Hirschsprung Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to investigate long term outcomes of surgical intervention for Hirschsprung's disease and to explore the relation between scintigraphic defecography, type of surgery performed and symptoms as evaluated by a disease specific questionnaire.

DETAILED DESCRIPTION:
Hirschsprung's disease (HD) is a congenital deficiency with incomplete development of nerves in the gastrointestinal tract leading to absence of peristalsis in the affected segment of bowel. Most patients require surgical intervention with removal of the affected segment of bowel. Physical symptoms affecting quality of life are not uncommon in patients born with HD in spite of surgical intervention. This renders a need for a tool for evaluating the functional outcome in these patients.

Scintigraphic defecography examines the defecation in terms of the ability to empty the bowel and examines the relocation of faeces within the bowel in relation to defecation.

This study aims to explore the relation between scintigraphic defecography, type of surgery performed and symptoms as evaluated by a disease specific questionnaire (Hirschsprung and Anorectal Malformations Quality of Life Questionnaire).

ELIGIBILITY:
Inclusion Criteria:

* Patients operated with any type of surgery for Hirschsprung's disease between 1985-2014
* Age > 15 years

Exclusion Criteria:

* Unable to understand given instructions in relation to the defecography (ex. retarded)
* Pregnancy
* Missing consent

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients operated for Hirschsprung's disease from 1985-2014 are gathered in a cohort, intended for several studies on Hirschsprung's disease. All patients > 15 years from this cohort will be invited to participate in this study.
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
Evacuation fraction (%) of radioactive material between first, second and third round of scintigraphic imaging | Day 1
  The fraction of evacuated radioactive material by defecation between rounds of scintigraphic imaging
Presence of retrograde movement of radioactive material (yes/no) | Day 1
  Presence of retrograde movement of radioactive material within the bowel on scintigraphic images between rounds of scintigraphic imaging
Hirschsprung and Anorectal Malformations Quality of life Questionnaire sub scales and total score | Day 1
  Disease specific questionnaire including sub scales for laxative and constipating diet, presence of diarrhoea and constipation, faecal and urinary incontinence, social and emotional functioning, body image, physical symptoms and sexual functioning. Each item is phrased as a multiple-choice question with four response options; never, once in a while, often and very often. Responses are linearly transformed on a 0-100 scale with a higher score indicating better QOL.
Type of surgical intervention performed in each individual (for example pull-through surgery) | Day 1
  Type of surgical intervention performed to treat Hirschsprung's disease

CONTACTS AND LOCATIONS:
Locations (1):
- Odense University Hospital, Odense, Region Syddanmark, Denmark